CLINICAL TRIAL: NCT01624181
Title: Identification of Microbes Through Detection of Pathogen Specific Volatile Compound Patterns, Using Multi-capillary Column Coupled Ion Mobility Spectrometry (MCC-IMS) in the Setting of Hospital-acquired Pneumonia
Brief Title: Fast Identification of Pathogen in the Setting of Hospital-acquired Pneumonia Using Ion Mobility Spectrometry
Status: Completed | Type: Observational
Sponsor: University of Göttingen (Other)
Collaborators: German Federal Ministry of Economics and Technology (Other Government); B&S Analytik GmbH, Dortmund, Germany (Unknown); Universität Duisburg-Essen (Other); Korean Institute for Science and Technology in Europe, Saarbrücken, Germany (Unknown)
Responsible Party: Principal Investigator, Dr. T. Perl, Principal Investigator, University of Göttingen
Other Study IDs: ZIM-KF2111207AK0; DRKS00004178 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2012-06-08; First posted 2012-06-20 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Acute Lower Respiratory Tract Infection; Pneumonia
Keywords: ion mobility spectrometry; hospital-acquired pneumonia; microbiological investigation; intensive care
MeSH Terms: conditions — Pneumonia; Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — aspiration samples from the respiratory system (tracheal secretion sample, BAL)
Oversight: Data Monitoring Committee: No

SUMMARY:
With this study the investigators want to determine, if a fast identification of germs, causing hospital-acquired infections of the lower respiratory tract, is possible through the use of MCC-IMS technology - a method that allows on time detection and identification of very small amounts of substances in gas samples. Therefore aspiration samples from the respiratory tracts of ventilated patients, which are suspected to develop such an infection, will be collected, cultivated and analyzed by MCC-IMS. The investigators want to determine if MCC-IMS diagnostic could be a faster alternative to conventional microbiological methods. The results of the MCC-IMS analyses therefore will be compared with results of conventional microbiological methods.

DETAILED DESCRIPTION:
In this clinical feasibility study it is to be investigated if MCC-IMS analyses over clinical samples from ventilated critically ill patients could be a fast and secure alternative to conventional microbiological diagnostic methods in the identification of human pathogenic microbes in the setting of hospital-acquired pneumonia. Therefore aspiration samples from intubated and ventilated critically ill patients, which are suspected to develop such an infection, will be collected and cultivated for a short period of time. The headspace over these cultures will be analyzed using MCC-IMS - a technology that allows on time detection and identification of very small amounts of substances in complex and humid gas samples. Conventional microbiological investigations, including MALDI-TOF, will be carried out parallel to the MCC-IMS analyses.

ELIGIBILITY:
Inclusion Criteria:

* patient is at the hospital for more than 48 hours
* patient is intubated and mechanically ventilated
* clinical suspicion for an infection of the lower respiratory tract has been raised and decision for microbiological investigation of respiratory aspirate was made

Exclusion Criteria:

* patient is at the hospital for less than 48 hours
* patient has been recruited for another clinical study
* suspicion for an infection with a germ belonging to risk class 3 and 4 according to the german law (BioStoffV and TRBA, e.g. Mycobacterium tuberculosis)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients will be recruited from two intensive care units of the university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Time until pathogen identification through MCC-IMS | Up to 24 hours after sampling. Sampling (as an iclusion criterion) can be necessary anytime along the ICU stay of the patient (up to 12 months).
  time from sampling until the availability of the results.
time until pathogen identification through conventional microbiological diagnostic methods | Up to 5 days after Sampling. Sampling (as an iclusion criterion) can be necessary anytime along the ICU stay of the patient (up to 12 months).
  time from sampling until the availability of the results.

SECONDARY OUTCOMES:
length of ICU stay | time from ICU admission to ICU discharge of study patients (up to 12 months)
  total LOS ICU
Type and dosage of administered antibiotic therapy | approximately 5 days. Starting with the day the samples are taken. Ending with the day on which the results microbiological test are made avaiable.
  name and dosage of the antibiotic therapeutic agents used to threat the infection
morbidity | Starts for study patients with the ICU admission and ends two days after the start of the initial antibiotic therapy. (up to 12 Months)
  morbidity of the critical ill patient at ICU admission, at the time of sampling and after two days of antibiotic therapy using the SAPS II scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Quintel, Prof. Dr., Study Director — University of Göttingen
Locations (1):
- University Medical Center Göttingen, Göttingen, Lower Saxony, Germany

REFERENCES:
- [Background] Junger M, Vautz W, Kuhns M, Hofmann L, Ulbricht S, Baumbach JI, Quintel M, Perl T. Ion mobility spectrometry for microbial volatile organic compounds: a new identification tool for human pathogenic bacteria. Appl Microbiol Biotechnol. 2012 Mar;93(6):2603-14. doi: 10.1007/s00253-012-3924-4. Epub 2012 Feb 12. PMID 22327321
- [Background] Perl T, Junger M, Vautz W, Nolte J, Kuhns M, Borg-von Zepelin M, Quintel M. Detection of characteristic metabolites of Aspergillus fumigatus and Candida species using ion mobility spectrometry-metabolic profiling by volatile organic compounds. Mycoses. 2011 Nov;54(6):e828-37. doi: 10.1111/j.1439-0507.2011.02037.x. Epub 2011 Jun 12. PMID 21668516